CLINICAL TRIAL: NCT07252557
Title: Effectiveness of Different Mouthwash Temperatures on Oral Mucositis Pain and Patient Comfort During Radiotherapy for Head and Neck Cancer: A Randomized Controlled Trial
Brief Title: Mouthwash Temperature and Oral Mucositis in Head and Neck Radiotherapy
Acronym: CoolRinseHNC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-CS2-25178
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer (H&Amp;Amp;N); Radiation-induced Oral Mucositis; Supportive Care; Nursing Interventions; Radiotherapy Side Effects
Keywords: Head and Neck Cancer; Radiation-Induced Oral Mucositis; Water Temperature; Cold Water Rinse; Supportive Care; Pain Management; Radiotherapy; Nursing Intervention
MeSH Terms: conditions — Head and Neck Neoplasms; Agnosia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Water Rinse (Experimental): Participants will rinse their mouth with cold water at approximately 15-20°C, four times daily for 30-60 seconds throughout six weeks of radiotherapy, followed by a two-week follow-up period.
  Interventions: Behavioral: Water Rinse at Different Temperatures
- Room Temperature Water Rinse (No Intervention): Participants will rinse their mouth with room-temperature water at approximately 30-35°C, with identical frequency and duration as the experimental arm.

INTERVENTIONS:
Behavioral: Water Rinse at Different Temperatures — rinse their mouth with cold water at approximately 15-20°C
  Arms: Cold Water Rinse

SUMMARY:
This single-center randomized controlled trial evaluates the effects of cold (15-20°C) versus room-temperature (30-35°C) water gargling on oral mucositis severity, pain, and comfort in patients with head and neck cancer undergoing radiotherapy. Participants will rinse their mouth four times daily for 30-60 seconds over a 6-week radiotherapy course, with follow-up for two additional weeks. The study hypothesizes that cold-water rinsing can reduce the severity of radiation-induced oral mucositis (RTOM) and pain, improve oral comfort, and minimize treatment interruptions.

DETAILED DESCRIPTION:
Radiation-induced oral mucositis (RTOM) is a frequent and debilitating side effect of radiotherapy for head and neck cancer, leading to pain, nutritional compromise, and potential treatment discontinuation. Cryotherapy and local temperature modulation have been proposed as low-cost, accessible nursing interventions that reduce inflammation through vasoconstriction and analgesia. This randomized trial will assess the clinical efficacy and patient acceptability of temperature-modulated water rinsing as a non-pharmacologic, supportive-care intervention. Subgroup analyses will examine differential responses among patients with dental sensitivity or betel-nut chewing habits.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed head and neck cancer (HNC) receiving radiotherapy for the first time, with or without concurrent chemotherapy.
* Conscious, communicative, and able to perform the rinsing procedure and complete questionnaires.
* Provided written informed consent prior to enrollment.

Exclusion Criteria:

* Non-HNC diagnoses or radiotherapy to sites outside the oral/oropharyngeal region.
* Cognitive impairment or inability to complete the rinsing protocol.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis Severity | Baseline (prior to radiotherapy), Week 2, Week 4, Week 6 (end of radiotherapy), and 2 weeks after completion of radiotherapy
  Assessed using WHO Oral Mucositis Grading Scale (0-4).
Pain Intensity (VAS 0-10) | Baseline (prior to radiotherapy), Weeks 1-6 during radiotherapy, and 2 weeks after completion of radiotherapy
  Patient-reported pain intensity using VAS (0-10).

SECONDARY OUTCOMES:
Oral Comfort | Baseline, Week 2, Week 4, Week 6 (end of radiotherapy)
  Assessed using a 5-point Likert comfort scale.
Satisfaction with Rinsing Modality | Week 6 (end of radiotherapy) and 2 weeks after completion of radiotherapy
  Satisfaction questionnaire evaluating acceptability of assigned water temperature.
Psychological Distress | Baseline (prior to radiotherapy) and Week 6 (end of radiotherapy)
  Psychological distress measured using the Brief Symptom Rating Scale (BSRS-5).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No